CLINICAL TRIAL: NCT02595086
Title: Multicenter Randomized Controlled Trial Comparing Laparoscopic Pylorus Preserving Gastrectomy Versus Laparoscopic Distal Gastrectomy for the Middle Third Early Gastric Cancer (KLASS-04)
Brief Title: Comparison of Laparoscopic Pylorus Preserving Gastrectomy Versus Laparoscopic Distal Gastrectomy
Acronym: KLASS-04
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KLASS-04
Record Dates: First submitted 2015-07-02; First posted 2015-11-03 (Estimated); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laparoscopic PPG (Experimental): Laparoscopy assisted pylorus-preserving gastrectomy(LPPG) with D1+ lymphadenectomy is performed (exclude lymph node station No. 5) in Japanese classification. Systemic en bloc lymph node dissection is mandatory. Resection margin should be negative for malignancy with intraoperative frozen biopsy. Extra-corporeal gastro-gastrostomy should be performed
  Interventions: Procedure: Laparoscopic PPG
- Laparoscopic DG (Active Comparator): Laparoscopic distal gastrectomy(LDG) with D1+ lymphadenectomy in Japanese classification. Systemic en bloc lymph node dissection is mandatory. Resection margin should be negative for malignancy with intraoperative frozen biopsy.
  Anastomosis method (extra-corporeal or intra-) and reconstruction type (Billroth I (gastroduodenostomy), Billroth II, or Roux-en Y gastrojejunostomy) are optional according to the surgeon's preference
  Interventions: Procedure: Laparoscopic DG

INTERVENTIONS:
Procedure: Laparoscopic PPG — Laparoscopy assisted pylorus-preserving gastrectomy with D1+ lymphadenectomy (exclude lymph node station No. 5) in Japanese classification.
  Arms: Laparoscopic PPG
Procedure: Laparoscopic DG — Laparoscopic distal gastrectomy with D1+ lymphadenectomy in Japanese classification.
  Arms: Laparoscopic DG

SUMMARY:
The aim of this study is to show better postoperative quality of life including lower incidence of dumping syndrome and comparable survival after laparoscopic pylorus preserving gastrectomy (LPPG), compared to laparoscopic distal gastrectomy (LDG) in patients with middle-third early gastric cancer

DETAILED DESCRIPTION:
Participating Surgeons

Prior to this clinical trial, only the surgeons who are considered to have the standardization by review committee participated.

Patients Registration

It is required to ensure that the patients meet the inclusion criteria for this clinical trial, are free from any items of exclusion criteria, are explained about the participation in the clinical trial along with the informed consent forms.

After rechecking the patients with the registration check list by accessing the web-based randomized program provided from Seoul National University Hospital Medical Research Collaborating Center.

Each group 128 patients, total 256 subjects will be enrolled.

Randomization

The registration randomization should be done with 1:1 ratio for each researcher.

Baseline number (BN) should be provided to the subjects in the order of acquisition of informed consent form. Based on the subjects who are selected as the appropriate subjects in the end, the allocation number (AN) shall be provided in the order of randomized allocation table.

Procedure

Operations are performed according to the allocated group.

ELIGIBILITY:
Inclusion Criteria:

Patients are included in the trial if they meet all of the following criteria:

* histologically proven primary gastric adenocarcinoma
* aged 20-80 years old
* performance status (PS) of 0 or 1 on Eastern Cooperative Oncology Group (ECOG) scale
* performance status (PS) of I to III on American Society of Anesthesiologists (ASA) score
* clinical stage T1N0M0, which are assessed by endoscopic ultrasound or computed tomography (CT) scan (AJCC 7th classification)
* location of primary tumor; middle third of stomach (more than 5cm away from the pylorus)
* written signed informed consent

Exclusion Criteria:

Patients are excluded if they meet any of the following criteria:

* pyloric deformity because peptic ulcer disease
* previous gastric surgery (e.g. gastro-jejunostomy, primary closure)
* synchronous lesion of early gastric cancer or adenoma in antrum
* prior treatment of endoscopic submucosal dissection, chemotherapy or radiation therapy against any other malignancies
* patients who need combined resection (eg. cholecystectomy)
* vulnerable patients (lack of decision-making capacity, pregnant, or breast-feeding women)
* participated in another clinical trial within the last six months or currently involved patients

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2015-07; Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dumping syndrome, assessed by Sigstad score (≥7) | 1 years postoperatively

SECONDARY OUTCOMES:
Relapse-free survival | 3 years postoperatively
Overall survival | 3 years postoperatively
Operative morbidity | 30 days for early morbidity
Operative mortality | mortality for 90 days
Body weight change | check at every visit up to 3 years postoperatively
Fat volume change on abdominal CT scan | check at every 1 year up to 3 years postoperatively
Change of Hemoglobin | check at every visit up to 3 years postoperatively
Change of Protein | check at every visit up to 3 years postoperatively
Change of Albumin | check at every visit up to 3 years postoperatively
QOL measurement (EORTC C30/STO22) (composite) | 6 month, 1 year, 2 year, 3 year postoperatively
Incidence of gallbladder stone | check at every 6 months up to 3 years postoperatively
Gross and microscopic changes measured by gastroscopy (composite) | 1 year, 2 year, 3 year postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Hyuk-Joon Lee, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (5):
- South Korea (5):
  - Kyungpook National University Hospital, Daegu, Jung-gu
  - National Cacner Center, Goyang-si
  - Department of Surgery, Seoul National University BUNDANG Hospital, Seongnam
  - Seoul National University Hospital, Seoul
  - Yonsei University Severance Hospital, Seoul

REFERENCES:
- [Derived] Park DJ, Kim YW, Yang HK, Ryu KW, Han SU, Kim HH, Hyung WJ, Park JH, Suh YS, Kwon OK, Yoon HM, Kim W, Park YK, Kong SH, Ahn SH, Lee HJ. Short-term outcomes of a multicentre randomized clinical trial comparing laparoscopic pylorus-preserving gastrectomy with laparoscopic distal gastrectomy for gastric cancer (the KLASS-04 trial). Br J Surg. 2021 Sep 27;108(9):1043-1049. doi: 10.1093/bjs/znab295. PMID 34487147